CLINICAL TRIAL: NCT07152054
Title: The Effect of Virtual Forest Bathing on Pain, Anxiety, Fear, Sleep Quality, Vital Signs, and Cortisol Levels in Patients Undergoing Bariatric Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Forest Bathing on Bariatric Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muazzez Merve TORAMAN, Research Assistant, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Muazzez TORAMAN
Record Dates: First submitted 2025-08-10; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Bariatric Surgery; Virtual Reality; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Virtual Forest Bathing (Experimental): Patients in the experimental group will undergo the routine surgical procedure implemented in the hospital, and their evaluations will be carried out using the predetermined questionnaires. In addition, they will receive a virtual forest bathing intervention on the evening prior to surgery and on the first postoperative day. On the day of admission for bariatric surgery, the researcher will administer, face-to-face, the Personal Information Form, Surgical Fear Questionnaire, Richard-Campbell Sleep Questionnaire, Visual Analog Scale (VAS) for pain assessment, State-Trait Anxiety Inventory, and the parameter recording form. Following the virtual forest bathing sessions conducted on the evening before surgery and on the first postoperative day, the Surgical Fear Questionnaire, Richard-Campbell Sleep Questionnaire, Visual Analog Scale (VAS), State-Trait Anxiety Inventory, and parameter recording form will be completed again.
  Interventions: Device: virtual forest bathing

INTERVENTIONS:
Device: virtual forest bathing — Virtual reality (VR) is an advanced computer technology and a novel technique used in healthcare to alleviate pain and provide patient comfort. It enables individuals to interact with a 360-degree virtual environment through a headset device. It has been observed that painful or emotionally stressful stimuli from the external world are diminished within the VR environment, with the individual's attention redirected and focused on this immersive setting.
  In our study, a 20-minute VR video will be used, providing the sensation of walking through a calming 360-degree virtual forest environment accompanied by natural sounds, viewed through VR headsets. Unlike some commercially available VR headsets, the Oculus Quest 2 model will be utilized, as it serves as both the computer and display system, eliminating the need for a smartphone. This device is preferred for its ability to deliver high-quality video without interruptions that might negatively affect the VR experience.
  After explaining

SUMMARY:
This study will be conducted at the General Surgery Clinic of City Hospital in Erzurum between August 2025 and April 2026 using a randomized controlled experimental design. In the power analysis, it was determined that the sample of the study should be 70 patients in total, 35 patients in each group, with a medium effect size of 0.5% according to Cohen (42), a margin of error of 0.05%, a confidence interval of 0.95%, and a 95% universe representation power. Patients will be assigned to either the experimental or control groups using a random number generator using a two-block randomization method (random.org). Given that exposure to nature through virtual reality increases physiological arousal and promotes positive mood, the study aimed to evaluate the effects of virtual forest bathing on pre- and postoperative pain, anxiety, fear, sleep, vital signs, and cortisol levels in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgery is considered an effective method for the treatment of obesity and is increasingly being performed worldwide. While bariatric surgery is an effective method for weight loss and control, the physiological changes caused by excess weight caused by surgical and anesthesia procedures can lead to postoperative complications. Before and after bariatric surgery, uncertainty about the surgical process, concerns about the surgical procedure and anesthesia procedures, and postoperative lifestyle changes and concerns about potential complications all contribute to an increased surgical stress response in obese individuals. Integrating non-pharmacological interventions into the treatment process, rather than focusing solely on pharmacological methods, is crucial. These approaches can be effective in alleviating the physical and psychological symptoms associated with surgery; they can support the recovery process by reducing anxiety and improving sleep quality. Techniques based on distraction, such as virtual reality, music therapy, and breathing exercises, do not produce any side effects, unlike pharmacological agents. These methods also help patients maintain basic physiological parameters such as blood pressure, respiration, and pulse rate, while also contributing to increased comfort and satisfaction. One of these innovative approaches is forest bathing, also known as "Shinrin-yoku," meaning "immersing in the forest atmosphere." Forest bathing utilizes the healing effects of forests to improve health and prevent disease through forest walks. Forest atmospheres are known to contain numerous healing factors that play an important role in the prevention and treatment of health problems through sensory input. There is evidence that forest bathing can help individuals regain attention and foster more positive emotions. Forest environments have positive effects on the cardiovascular system, nervous system, endocrine system, immune system, and mental health. This study was designed considering the need for evidence regarding the pre- and postoperative use of virtual forest bathing in the context of nursing care. It is believed that virtual forest bathing may have positive effects on pain, anxiety, fear, sleep patterns, cortisol, and vital signs in patients undergoing bariatric surgery during the pre- and postoperative periods. Virtual forest bathing has demonstrated successful results in various areas and with different patient groups for reducing stress and anxiety. However, there are limited studies specifically related to bariatric surgery, both in our country and elsewhere. Some studies abroad have shown that such psychological support methods have positive effects on surgical stress, but the number of studies conducted in this area in our country is quite limited. Therefore, this study is valuable in providing scientific data to healthcare professionals in our country. As experimental research on forest bathing intensifies, medical and healthcare professionals have focused on the forest's ability to boost immunity and reduce stress. They have concluded that even short-term forest bathing can help strengthen the body's immune system and improve mood. Implementing holistic, non-pharmacological interventions for patients experiencing both physical and psychological challenges before and after bariatric surgery is crucial. Virtual reality-based nature interventions are considered among the innovative and effective approaches that can be integrated into nursing care during this process. In this context, the study aimed to evaluate the effects of virtual forest bathing on pain, anxiety, fear, sleep patterns, vital signs, and cortisol in patients undergoing bariatric surgery before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Ability to communicate verbally
* Absence of any psychiatric disorder
* Undergoing bariatric surgery
* No prior experience with virtual forest bathing

Exclusion Criteria:

* Inability to establish communication
* Presence of major hearing or visual impairment
* Presence of any condition that may affect decision-making ability (e.g., psychological disorders, dementia)
* Use of medications that may affect cognitive status (e.g., sedatives, antipsychotics)
* Patients who report having previously experienced virtual forest bathing will be excluded from the sample

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form: | up to 24 hours
  This questionnaire, developed by the researcher based on a literature review related to the topic, consists of 16 questions addressing variables such as gender, age, education level, marital status, and previous surgical history.
Surgical Fear Questionnaire (SFQ) | up to 24 hours
  Surgical Fear Questionnaire (SFQ):
  Developed by Theunissen et al. in 2014 to assess the fear levels of patients scheduled for surgical procedures, this 8-item Likert-type scale evaluates short-term surgical fears with items 1-4 and long-term surgical fears with items 5-8. Each item is scored on a scale from 0 ("not afraid at all") to 10 ("very afraid"), resulting in a total score ranging from 0 to 80. Higher scores indicate greater levels of surgical fear (Theunissen et al., 2014). The Turkish validity and reliability study conducted by Bağdigen and Özlü (2018) reported a Cronbach's alpha coefficient of 0.93.
Richard-Campbell Sleep Questionnaire (RCSQ) | up to 24 hours
  Developed by Richards in 1987 (Richards, 1987) and adapted into Turkish by Özlü and Özer in 2015 (Özlü & Özer, 2015), this scale consists of six items evaluating sleep depth, time to fall asleep, frequency of awakenings, time to return to sleep after awakening, sleep quality, and environmental noise level. Each item is scored between 0 and 100. In total score calculation, the sixth item (noise level) is excluded, and scoring is based on the remaining five items. Higher scores indicate better sleep quality. Final scores are calculated by dividing the total score by the number of items. Scores between 0-25 indicate "very poor" sleep quality, while scores between 76-100 indicate "very good" sleep quality.
Visual Analog Scale (VAS) | up to 24 hours
  Developed by Price et al. (1983), this scale measures the intensity of pain using a 10 cm vertical or horizontal line with endpoints labeled as "no pain" (0) and "worst possible pain" (10). The patient marks a point corresponding to their perceived pain intensity, and the distance from the "no pain" end to the marked point is measured in centimeters, representing the pain score. Higher scores indicate greater pain intensity.
State-Trait Anxiety Inventory (STAI-STAII) | up to 24 hours
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Oner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Tracking Form for Parameters | up to 24 hours
  Before and after bariatric surgery, patients' heart rate, blood pressure, and oxygen saturation will be measured and recorded in this form. In addition, to assess stress levels, blood cortisol measurements will be performed. Blood samples for cortisol will be collected in the morning (between 07:30-08:30) in appropriate tubes, promptly transported to the laboratory, and analyzed under cold chain conditions. Serum or plasma will be separated and analyzed using standard devices. All procedures will be carried out in the Erzurum City Hospital laboratory according to existing standard protocols and high-quality criteria, and results will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Muazzez Merve TORAMAN, Principal Investigator — Atatürk Üniversity

IPD SHARING:
Plan to Share IPD: No